CLINICAL TRIAL: NCT02151461
Title: A Randomized, Double-Blind, Active-Controlled Study to Evaluate the Effect of Various Fixed-Dose Leucine and Metformin Combinations (NS-0100) Versus Standard Metformin Monotherapy on Glycemic Control in Subjects With Type 2 Diabetes
Brief Title: Dose Comparisons of Leucine-Metformin Combinations on Blood Glucose Levels In Type 2 Diabetic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NuSirt Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NS-0100-01
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Metformin; Leucine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low Metformin (Experimental): 3 capsules BID with each capsule containing 366.7 mg L-Leucine and 41.7 mg of metformin
  Interventions: Drug: Low Metformin
- Mid Metformin (Experimental): 3 capsules BID with each capsule containing 366.7 mg L-Leucine and 83.3 mg of metformin
  Interventions: Drug: Mid Metformin
- High Metformin (Experimental): 3 capsules BID with each capsule containing 366.7 mg L-Leucine and 166.7 mg of metformin
  Interventions: Drug: High Metformin
- Metformin Monotherapy (Experimental): 3 Capsules BID each containing 166.7 mg of metformin with dose escalation to 283.3 mg capsules BID (1,700 mg/Day) at Day 14.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Low Metformin — 1100 mg L Leucine in combination with 125 mg of Metformin BID
  Other Names: Metformin; Leucine; L-Leucine
  Arms: Low Metformin
Drug: Metformin — 500 mg metformin BID until day 14 with dose escalation at day 14 to 850 mg metformin BID
  Arms: Metformin Monotherapy
Drug: Mid Metformin — 1100 mg of Leucine in combination with 250 mg Metformin BID
  Other Names: Metformin; Leucine; L-Leucine
  Arms: Mid Metformin
Drug: High Metformin — 1100 mg of Leucine in combination with 500 mg Metformin BID
  Other Names: Metformin; Leucine; L-Leucine
  Arms: High Metformin

SUMMARY:
The goal of this study is to demonstrate that leucine in combination with a low does of metformin can serve as an adjunct to diet and exercise to improve blood glucose levels in type 2 diabetic subjects. This study will compare three doses of a leucine-metformin combination to the standard metformin dose in controlling blood glucose levels in type 2 diabetic patients.

DETAILED DESCRIPTION:
This is a randomized, 4-week, active-controlled, double-blind study to evaluate the effect of various fixed-dose combinations of leucine and metformin compared to standard metformin monotherapy on glycemic control. In this study, standard metformin therapy will be defined as 1000 g/day for Day 1 to Day 14 and then escalated to 1700 g/day for Day 15 to Day 28. Subjects meeting all inclusion criteria and no exclusion criteria will be randomized to one of four treatment arms.

The primary objective of the study is to evaluate the change in fasting plasma glucose from Baseline (Day 1) to Week 4 (Day 28) in subjects receiving various fixed-dose combinations of leucine and metformin compared to standard metformin monotherapy. Secondary objectives will also assess changes in baseline-corrected plasma glucose and insulin area under the concentration curves from baseline to day 28 and changes in insulin secretory rates as assessed during a 3-hour meal tolerance test. Finally the effects of gastrointestinal symptoms will be assessed by subject questionnaires.

The study will include a total of 3 periods: screening or washout of current diabetic monotherapy, a pre-treatment period to ensure subjects will be compliant, and a treatment period of 4 weeks, with the first dosing of medication on day 1 of the study. Each day blood glucose readings will be measured and recorded by patients. Three-hour standardized meal tests will be performed at Baseline (Day 1) and at Study Termination (Day 28). In addition, two, 7-day continuous glucose assessments will be conducted, as well as two seven point glucose profiles. Patients will also be asked about any gastrointestinal side effects they experience.

ELIGIBILITY:
Inclusion Criteria:

* Over age 18 at study entry.
* Male, or female, if female, meets all of the following criteria:
* Not breastfeeding
* Post-menopausal or negative pregnancy test result (human chorionic gonadotropin, beta subunit [β- hCG]) at Screening (Visit 1) (not required for hysterectomized females)
* If of childbearing potential and sexually active, must practice and be willing to continue to practice appropriate birth control
* Is diagnosed with type 2 diabetes mellitus and either not adequately controlled by: diet and exercise alone or diet and exercise plus a single, first line treatment for type 2 diabetes.
* If treated with an oral anti-diabetes agent, be willing and able to withdraw from therapy for 4 weeks after the screening visit and prior to initiating study mediation at Baseline (Day 1/Visit 4).
* Be willing to avoid acetaminophen use for intervals up to 10 days as required for study procedures (see Section 4.6)
* Has a fasting plasma glucose ≥126 mg/dL to ≤220 mg/dL at Screening
* Has an HbA1c ≥7% to ≤8.5% at Screening
* Has a BMI ≤40 kg/m2
* Clinical laboratory tests (hematology, clinical chemistry, and urinalysis) either normal or abnormal but consistent with type 2 diabetes mellitus.
* Is able to read, understand, and sign the informed consent forms (ICF) and if applicable, an authorization to use and disclose protected health information form (consistent with health insurance portability and accountability act of 1996 [HIPAA] legislation), communicate with the investigator, and understand and comply with protocol requirements.

Exclusion Criteria:

* Clinically significant renal dysfunction
* If using any of the following medications, has not been on a stable treatment regimen for a minimum of 4 weeks prior to screening:

Lipid-lowering agents Anti-hypertensive medications Thyroid replacement therapy Non-steroidal anti-inflammatory agents

* Unable to perform self-blood glucose monitoring employing a glucose meter.
* History of active cardio- or cerebro-vascular disease with an event within the previous 6 months
* Gastrointestinal disorders
* Endocrine disorders other than type 2 diabetes
* Chronic infection
* Hepatic disease
* Neurological or psychiatric diseases
* History of other psychiatric disorders
* Has been treated (within the last month), is currently treated, or is expected to require or undergo treatment with; any anti-diabetes medications (other than as allowed by the inclusion criteria), oral or parenteral steroids.
* Participation in a weight loss program within the past 3 months.
* Weight change by more than 10 pounds during the past month.
* History of alcohol or substance abuse in the past 3 months or a positive screen for alcohol or drugs of abuse at screening.
* Has received any investigational drug within 3 months of Screening.
* Has donated blood within 3 months before Screening or is planning to donate blood during the study.
* Has known allergies or hypersensitivity to metformin or leucine
* Is employed, contracted or has an immediate family member directly affiliated with NuSirt Biopharma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orville G Kolterman, MD, Study Chair — NuSirt Biopharma
Locations (9):
- United States (9):
  - Catalina Research Institute, Chino, California
  - Palm Beach Research, Palm Beach, Florida
  - Meridien Research, Tampa, Florida
  - River Birch Research Alliance, Blue Ridge, Georgia
  - Meridian Research, Savannah, Georgia
  - Streling Research Group, Cincinnati, Ohio
  - Medical Research South, Charleston, South Carolina
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University Medical Center, Diabetes, Endocrinology, and Metabolism, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects meeting all inclusion criteria and no exclusion criteria were randomized to one of four treatment arms in the ratio of 1:1:1:1 (A:B:C:D). The randomization was stratified by fasting plasma glucose (≥126 mg/dL to <200 mg/dL, and ≥200 mg/dL to ≤220 mg/dL), as well as metformin experience. Yes/No history of abdominal side effects.
Groups:
- FDC125: Leucine 1100mg +Metformin 125mg
- FDC250: Leucine 1100mg +Metformin 250mg
- FDC500: Leucine 1100mg +Metformin 500mg
- Control: Day 1-14: 500mg, Day 15-28: 850mg
Period: Overall Study
Arm/Group | FDC125 | FDC250 | FDC500 | Control
Started | 24 | 25 | 24 | 23
Completed | 18 | 24 | 21 | 19
Not Completed | 6 | 1 | 3 | 4
Not completed — Adverse Event | 5 | 1 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1
Not completed — Treatment discontinuation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who had adequate exposure to the randomized study medication during the 4-week treatment period (Day 1/Visit 4 to Day 28/Visit 7) and had adequately complied with the protocol as assessed by the sponsor prior to database lock.The groups in Metformin experience are mutually exclusive.
Groups:
- Total: Total of all reporting groups
Arm/Group | FDC125 | FDC250 | FDC500 | Control | Total
Number analyzed (Participants) | 24 | 25 | 24 | 23 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] — Subjects who met the inclusion criteria, with FPG>126 to <220 mg/dL, HbA1c>7 to<8.5% and BMI<40kgm2
  years | 53.6 (9.87) | 55.1 (8.3) | 56.1 (10.08) | 59.3 (9.64) | 56.0 (9.56)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 19 | 21 | 18 | 17 | 75
  ≥65 years | 5 | 4 | 6 | 6 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 13 | 10 | 51
  Male | 9 | 12 | 11 | 13 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 15 | 12 | 12 | 53
  Not Hispanic or Latino | 10 | 10 | 12 | 11 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 5 | 6 | 16
  White | 22 | 20 | 19 | 16 | 77
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 87.049 (17.3747) | 88.584 (19.4687) | 84.493 (19.8622) | 86.777 (16.5700) | 86.745 (18.1696)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.142 (4.7113) | 30.985 (5.5766) | 29.927 (5.1504) | 31.146 (4.5838) | 30.798 (4.9778)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 194.3 (50.86) | 170.3 (44.28) | 182.8 (40.97) | 184.7 (50.87) | 182.9 (46.93)
Haemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: %] | 7.95 (0.837) | 8.01 (0.713) | 7.82 (0.563) | 8.24 (0.831) | 8.00 (0.747)
Previous Metformin experience [Count of Participants; unit: Participants]
  No Previous Experience | 4 | 1 | 5 | 3 | 13
  No Abdominal side effects from prior Metformin | 18 | 20 | 17 | 16 | 71
  Had Abdominal side effects from prior Metformin | 2 | 4 | 2 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 28 in Absolute Plasma Glucose Area Under the Curve (AUC) 0-3hr
Description: The primary endpoint for NS 0100 01 was the absolute plasma glucose AUC (0-3 hr) change from Day 1 to Day 28.
Time Frame: 0, 15min, 30min, 45min, 1hr, 1.5hrs, 2hrs, 2.5hrs and 3 hrs
Population: Mixed Model Inferential Statistical Analysis of Plasma Glucose AUC change from day 1-day 28 Evaluable Population (n=73)
Measure: Mean (Standard Deviation); unit: mg*hrs/dL
Arm/Group | FDC125 | FDC250 | FDC500 | Control
Number analyzed (Participants) | 17 | 18 | 20 | 18
mg*hrs/dL | -18.005 (142.8374) | -45.029 (114.6701) | -64.010 (146.0917) | -141.848 (194.9300)
Statistical Analysis 1: Comparison: FDC125 vs Control; Test type: Other — A mixed-effects model for analysis of covariance (ANCOVA) was used to analyze changes from Baseline in plasma glucose AUC(0-3hr) at Week 4 in the Day 28 Evaluable population. The model includes factors for treatment group and fasting plasma glucose stratum; p = 0.0435, ANCOVA — Baseline plasma glucose AUC(0-3hr) is adjusted as a covariate
Statistical Analysis 2: Comparison: FDC250 vs Control; Test type: Other; p = 0.065, ANCOVA
Statistical Analysis 3: Comparison: FDC500 vs Control; Test type: Other; p = 0.1216, ANCOVA

2. Secondary Outcome: Change From Baseline to Day 28 in Incremental Plasma Glucose Area Under the Curve (AUC)
Description: The baseline incremental (baseline-subtracted) glucose AUC0-3h was evaluated for treatment differences at baseline.
Time Frame: Baseline, Day 28
Population: Mixed Model Inferential Statistical Analysis of Incremental Plasma Glucose AUC change from day 1-day 28 Evaluable Population (n=73)
Measure: Mean (Standard Deviation); unit: mg*hrs/dL
Arm/Group | FDC125 | FDC250 | FDC500 | Control
Number analyzed (Participants) | 17 | 18 | 20 | 18
mg*hrs/dL | -2.338 (60.2834) | -17.614 (93.1243) | -23.061 (64.6290) | -29.604 (86.1126)
Statistical Analysis 1: Comparison: FDC125 vs Control; Test type: Other — A mixed-effects model for analysis of covariance (ANCOVA) was used to analyze changes from Baseline in incremental plasma glucose AUC at Week 4 in the Day 28 Evaluable population. The model will include factors for treatment group and fasting plasma glucose stratum; p = 0.8867, ANCOVA; The model includes factors for treatment group and fasting plasma glucose stratum
Statistical Analysis 2: Comparison: FDC250 vs Control; Test type: Other; p = 0.7641, ANCOVA
Statistical Analysis 3: Comparison: FDC500 vs Control; Test type: Other; p = 0.2518, ANCOVA

3. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change in fasting plasma glucose for the fixed dose leucine and metformin combination treatments A, B and C was evaluated.
Time Frame: Baseline, Day 28
Population: Mixed Model Inferential Statistical Analysis of Fasting Plasma Glucose change from day 1-day 28 Evaluable Population (n=73)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | FDC125 | FDC250 | FDC500 | Control
Number analyzed (Participants) | 17 | 18 | 20 | 18
mg/dL | -6.8 (36.91) | -9.7 (26.50) | -13.4 (38.55) | -36.0 (47.36)
Statistical Analysis 1: Comparison: FDC125 vs Control; Test type: Other; p = 0.0179, ANCOVA; Total daily dose is twice the respective dose, Pairwise comparison using Treatment D as the reference group
Statistical Analysis 2: Comparison: FDC250 vs Control; Test type: Other; p = 0.0736, ANCOVA
Statistical Analysis 3: Comparison: FDC500 vs Control; Test type: Other; p = 0.0475, ANCOVA

4. Secondary Outcome: Change in Hemoglobin A1c (HbA1c)
Description: Changes in HbA1c which is a marker of long-term glucose control was assessed.
Time Frame: Baseline, Day 28
Population: Mixed Model Inferential Statistical Analysis of HbA1c change from day 1-day 28 Evaluable Population (n=73)
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | FDC125 | FDC250 | FDC500 | Control
Number analyzed (Participants) | 17 | 18 | 20 | 18
percent | 0.11 (0.448) | -0.16 (0.485) | -0.01 (0.442) | -0.23 (0.607)
Statistical Analysis 1: Comparison: FDC125 vs Control; Test type: Other; p = 0.0089, ANCOVA; Total daily dose is twice the respective dose. Pairwise Comparison using Treatment D as the Reference Group
Statistical Analysis 2: Comparison: FDC250 vs Control; Test type: Other; p = 0.376, ANCOVA
Statistical Analysis 3: Comparison: FDC500 vs Control; Test type: Other; p = 0.0578, ANCOVA

5. Secondary Outcome: Change in Homeostasis Model Assessment-estimated Insulin Resistance (HOMA-IR)
Description: Effect on insulin sensitivity across fixed-dose leucine and metformin combination treatments or the standard metformin reference treatment.
Time Frame: Baseline, Day 28
Population: Mixed Model Inferential Statistical Analysis of HOMA-IR. Some of the samples collected were not viable and could not be included in the analysis. So, the total samples collected were still the same but since they could not be included in the analysis the exact number analyzed is referenced.
Measure: Mean (Standard Deviation); unit: HOMA units
Arm/Group | FDC125 | FDC250 | FDC500 | Control
Number analyzed (Participants) | 17 | 18 | 17 | 16
HOMA units | -0.31 (1.010) | -0.14 (0.548) | 0.11 (0.958) | -0.18 (1.017)
Statistical Analysis 1: Comparison: FDC125 vs Control; The HOMA Calculator,is an algorithm that takes account of variations in hepatic and peripheral glucose resistance, increases in insulin secretion curve for plasma glucose concentrations above 10 mmol/L (180 mg/dL), and contribution of circulating proinsulin (eg, C-peptide) to estimate steady state beta cell function (%HOMA-B) and insulin sensitivity (%HOMA-S), as percentages of a normal reference population. %HOMA-IR was analyzed on a logarithmic scale (natural logarithmic transformation); Test type: Other; p = 0.2177, ANCOVA; Total daily dose is twice the respective dose. Pairwise Comparison using Treatment D as the Reference Group
Statistical Analysis 2: Comparison: FDC250 vs Control; Test type: Other; p = 0.4144, ANCOVA
Statistical Analysis 3: Comparison: FDC500 vs Control; Test type: Other; p = 0.3117, ANCOVA

6. Secondary Outcome: Change In 7-Point Glucose Profiles
Description: The meal induced glucose change in pre-meal and post-meal glucose were measured 7 times during the day. Subjects self-monitored blood glucose (preprandial and postprandial) concentrations at least 7 times, including before and 1 to 2 hours after breakfast, lunch, dinner, and snacks). For each study day, the pre-meal values from the 7 point test for each subject were averaged to generate a single pre-meal glucose value. Similarly, for each study day the post-meal values from the 7-point test for each subject were averaged to generate a single post-meal glucose value. The average change from baseline (i.e., [(Mean Pre/Post-meal value at Day 28 - Mean Pre/Post-meal value at Baseline) + (Mean Pre/Post-meal value at Day 21- Mean Pre/Post-meal value at Baseline) + (Mean Pre/Post-meal value at Day 7- Mean Pre/Post-meal value at Baseline)]/ 3) over multiple time points listed in Time Frame. The mean pre-meal and post-meal values for baseline, day7, day 21 and day28 were used for comparison.
Time Frame: Baseline, Day 7, Day 21, Day 28
Population: Mixed Model Inferential Statistical Analysis of 7 point glucose change from day 1-day 28 Evaluable Population (n=73). Some of the samples collected were not viable and could not be included in the analysis. The total samples collected were still the same but since they could not be included in the analysis the exact number analyzed is referenced.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | FDC125 | FDC250 | FDC500 | Control
Number analyzed (Participants) | 16 | 17 | 18 | 15
mg/dL
  28 day change in Pre-meal Glucose Level | -6.50 (32.343) | -8.96 (61.561) | -25.51 (42.198) | -53.78 (45.488)
  28 day change in Post-meal Glucose Level | -15.98 (33.966) | 10.56 (44.944) | -34.25 (77.268) | -50.33 (60.756)
Statistical Analysis 1: Comparison: FDC125 vs Control; Test type: Other — Average Change in Pre-meal Glucose Level; p = 0.011, ANCOVA; Total daily dose is twice the respective dose Pairwise comparison using Treatment D as the reference group
Statistical Analysis 2: Comparison: FDC250 vs Control; Test type: Other — Average Change in Pre-meal Glucose Level; p = 0.0152, ANCOVA
Statistical Analysis 3: Comparison: FDC500 vs Control; Test type: Other — Average Change in Pre-meal Glucose Level; p = 0.0284, ANCOVA
Statistical Analysis 4: Comparison: FDC125 vs Control; Test type: Other — Average Change in Post-meal Glucose Level; p = 0.1273, ANCOVA; Total daily dose is twice the respective dose Pairwise comparison using Treatment D as the reference group
Statistical Analysis 5: Comparison: FDC250 vs Control; Test type: Other — Average Change in Post-meal Glucose Level; p = 0.0085, ANCOVA
Statistical Analysis 6: Comparison: FDC500 vs Control; Test type: Other — Average Change in Post-meal Glucose Level; p = 0.1289, ANCOVA

7. Secondary Outcome: Plasma Insulin Absolute and Incremental Meal Tolerance Test Area Under the Curve (AUC) 0-2hr
Description: Change in meal tolerance test insulin area under the curve (0-2 hr) from Day 1 to Day 28 for fixed-dose leucine and metformin combination treatments.
Time Frame: Baseline,Day 28
Population: Mixed Model Inferential Statistical Analysis of Plasma Insulin AUC and Incremental AUC change from day 1-day 28 Evaluable Population (n=73). Some samples collected were not viable. The total samples collected were still the same but since they couldn't included in the analysis, exact number analyzed is referenced.
Measure: Mean (Standard Deviation); unit: h*ulU/ml
Arm/Group | FDC125 | FDC250 | FDC500 | Control
Number analyzed (Participants) | 17 | 18 | 19 | 17
h*ulU/ml
  Plasma Insulin Absolute | -0.19 (74.531) | -5.64 (31.360) | -9.59 (34.987) | -18.06 (35.473)
  Plasma Insulin Incremental | 4.18 (67.120) | -4.25 (29.514) | -9.99 (27.956) | -15.91 (26.720)
Statistical Analysis 1: Comparison: FDC125 vs Control; Test type: Other — Plasma Insulin Absolute AUC(0-2hr) (h*uIU/mL); p = 0.3143, ANCOVA; Total daily dose is twice the respective dose. Pairwise comparison using Treatment D as the reference group
Statistical Analysis 2: Comparison: FDC250 vs Control; Test type: Other — Plasma Insulin Absolute AUC(0-2hr) (h*uIU/mL); p = 0.5677, ANCOVA
Statistical Analysis 3: Comparison: FDC500 vs Control; Test type: Other — Plasma Insulin Absolute AUC(0-2hr) (h*uIU/mL); p = 0.8407, ANCOVA

8. Secondary Outcome: Change From Baseline to Day 28 in Fasting Plasma Insulin Concentration
Description: Effect on fasting plasma insulin concentrations across fixed-dose leucine and metformin combination treatments or the standard metformin reference treatment was evaluated.
Time Frame: Baseline, Day 28
Population: Mixed Model Inferential Statistical Analysis of Plasma Insulin AUC and Incremental AUC change from day 1-day 28 Evaluable Population (n=73). Some collected were not viable. So, the total samples collected were still the same but since they could not be included in the analysis the exact number analyzed is referenced.
Measure: Mean (Standard Deviation); unit: h*uIU/mL
Arm/Group | FDC125 | FDC250 | FDC500 | Control
Number analyzed (Participants) | 17 | 18 | 19 | 17
h*uIU/mL | -2.06 (6.652) | -0.74 (4.069) | 0.20 (7.278) | -1.03 (7.694)
Statistical Analysis 1: Comparison: FDC125 vs Control; Test type: Other; p = 0.9789, ANCOVA; Total daily dose is twice the respective dose Pairwise comparison using Treatment D as the reference group
Statistical Analysis 2: Comparison: FDC250 vs Control; Test type: Other; p = 0.841, ANCOVA
Statistical Analysis 3: Comparison: FDC500 vs Control; Test type: Other; p = 0.748, ANCOVA

ADVERSE EVENTS:
Time Frame: 30 days
Description: Treatment-Energent Adverse Event (TEAE) is defined as an adverse event occurring on or after the first dose of randomized study medication, or existing prior to the time of and worsening after the time of the first dose of randomized study medication. Subjects experiencing multiple episodes of a given adverse event are counted once. This was a 28 day study and adverse event reporting went upto day 30.
Arm/Group | FDC125 | FDC250 | FDC500 | Control
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25 | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/24 | 1/25 | 0/24 | 1/23
Other Adverse Events (participants affected / at risk) | 3/24 | 3/25 | 3/24 | 5/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FDC125 (N=24) | FDC250 (N=25) | FDC500 (N=24) | Control (N=23)
Lacunar Infarction (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FDC125 (N=24) | FDC250 (N=25) | FDC500 (N=24) | Control (N=23)
Gastric Disorders (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2) | 5 (5)
Infections (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Food (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Nervous Disorders (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Respiratory Disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Abdominal Distension (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperglycemia (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes